CLINICAL TRIAL: NCT06385041
Title: Impact of Interactive Physical Therapy for Functional Capacity, Fear of Falls, Motivation and Quality of Life After Open Heart Surgery Due to Ischemic Heart Disease and Frailty in the Second Stage of Rehabilitation.
Brief Title: Cardiac Rehabilitation and Frailty Physical Training Program in Elderly Patients After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitalija Stonkuvienė (Other)
Responsible Party: Sponsor-Investigator, Vitalija Stonkuvienė, Principal Investigator, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BE-2-83
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Frailty; Surgery
Keywords: frailty syndrome; open heart surgery; cardiac rehabilitation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Physical training program will include: dosed aerobic training program on cycle ergometers (6 days/week, for 10-30 minutes, 30-50% watts or 30-50% HRmax). The training program consists individually according to the person state of health and respiratory muscle training (7 days/week, for 15 minutes).
- Multicomponent training group (Experimental): Physical training program will include: dosed aerobic training program on cycle ergometers and respiratory muscle trainings as in control group. Also patients will get an individualized exercise program for frailty syndrome, which will include strength exercises (with elastic resistance bands and weights) and balance training (unstable surfaces) 3 times/week 30-45 minutes.
  Interventions: Other: Multicomponent training group
- Computer-based interactive training group (Experimental): Physical training program will include: dosed aerobic training program on cycle ergometers and respiratory muscle trainings as in control group. Also patients will get an individualized program for frailty syndrome, with the help of interactive technologies 3 times/week. 30-45 minutes (gait training with Biodex GaitTrainerTM3 with visual and audio feedback, Zebris FDM-T, with the help of which virtual barriers are created, thus simulating real environment for the patient, while performing a cognitive task, for balance training investigators used a computerized Biodex board. For strength training investigators used equipment HUR based on pneumatic (air pressure) technology.
  Interventions: Other: Computer-based interactive training group

INTERVENTIONS:
Other: Multicomponent training group — Additional exercise program with balance and strength trainings will include 3 times/week. Patients will get an individualized exercise program for frailty syndrome, which will include strength exercises (with elastic resistance bands and weights up to 2kg 30-50% 1RM) and balance training (with unstable surfaces). The program will be performed by 3 sets with 10 repetitions 3 times/week 30-45 minutes.
  Arms: Multicomponent training group
Other: Computer-based interactive training group — Additional exercise program with balance and strength trainings will include 3 times/week 30-45 minutes. Patients will get an individualized program for frailty syndrome, with interactive technologies: gait training with Biodex GaitTrainerTM3 with visual, audio feedback and incline up to 10-15 min, Zebris FDM-T, with virtual barriers, thus simulating real environment for the patient, while performing a cognitive task up to 10-15 min, for balance training investigators used a computerized Biodex board. Exercises will be performed with the programs: Postural stability training, Limits of stability training, Weight shift training, Maze control training, Random control training, Percent weight-bearing training. For strength training investigators used equipment HUR based on pneumatic (air pressure) technology. For strength training intensity 30-50% 1-RM, 10 repetitions with 3 sets. Leg press, leg extension, leg abduction, leg adduction will be performed with pneumatic technology.
  Arms: Computer-based interactive training group

SUMMARY:
The aim of the research - to evaluate the impact of interactive physical therapy tools for functional capacity, fear of falls, motivation and quality of life after open heart surgery due to ischemic heart disease and frailty in the second stage of rehabilitation.

DETAILED DESCRIPTION:
The clinical trial will be performed during patient rehabilitation. All examination of the patient will be performed before rehabilitation and at the end of rehabilitation. Total subjects will spend 20 days in rehabilitation. All subjects who will have frailty syndrome will be assigned to one of three groups: control, intervention group-1 or intervention group-2.

ELIGIBILITY:
Inclusion Criteria:

* Patient's agreement to participate in the study,
* Age 65 years and older,
* Patients admitted to cardiac rehabilitation after open heart surgery,
* Patients with frailty (Edmonton frailty scale ≥4)
* 6-minute walk distance (6-MWD) ≥150 meters and walking without mobility aid.

Exclusion Criteria:

* Patient's disagreement to participate in the study
* Exercise-limiting comorbidities (primarily orthopedic and neurological conditions that would exclude individuals from participating in cardiac rehabilitation according to study protocol), cognitive, vision, linguistic deficits, chronic heart failure Class IV, anemia, wound healing disturbance or other various acute conditions that may limit active participation in physical therapy programs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Collecting data from the medical history | baseline
  comorbidities, date of surgery, etc. only with the subject's agreement
Frailty level by Edmonton frail scale score | baseline
  The Edmonton frail scale assesses 9 domains: cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance. Frailty level is measured by the Edmonton frail scale score - 0-3 - fit, 4-5 - vulnerable, 6-7 - mild frailty, 8-9 - moderate frailty,10-17 - severe frailty.
Fear of Falling by Falls Efficacy Scale International; FES-I). | baseline, 20 days.
  The FES-1 was used to assess the fear of falling level of participants about falling during indoor or outdoor activities. It has 16 items scored on a four-point Likert scale. assess the fear of falling level of participants about falling during indoor or outdoor activities minimum score 16 maximum score 64. The level of concern for each item is scored on a 4-point scale (1: not at all, 2: somewhat, 3: quite a lot, 4: very), with the total score range being 16 to 64.The results are divided into 3 parts: low 16-19, moderate 20-27, and high concern 28-64 points.
Quality of life by EuroQoL FiveDimensionsEQ-5D-5L. | baseline, 20 days.
  The EQ-5D-5L consists of 2 parts: descriptive system and visual analogue scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS (visual analogue scale) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Motivation by Multidimensional Health Locus of Control scale | baseline, 20 days.
  It is one of the most commonly-used parameters of health belief in planning the health education programs. The health locus of control is the degree to which individual believe that his or her behavior is controlled by external or internal factors. The survey contains with 18 items and consist of three subscales, namely Internal Health Locus of Control, Powerful Others Health Locus of Control, and Chance Health Locus of Control. Each of these subscales contains six items with a six-point Likert response scale ranging from 'Strongly Agree' to 'Strongly Disagree'. Scores for each subscale reflect the total score for the corresponding 6 items, with subscales having a minimum score of 6 and maximum score of 36.
Change from baseline functional capacity by six minutes walking test (6MWT) | baseline, 20 days.
  6MWT measured by meters. This test is performed preferably indoors, on a flat, straight,hard-surfaced corridor usually at least 30m long. The patient is told to be wear comfortable clothing and shoes. The physical therapist records heart rate and brachial arterial blood pressure and the Borg scale rating for dyspnea and fatigue before and after the test.
Change from baseline physical performance by Short Physical Performance Battery (SPPB) | baseline, 20 days.
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests.The scores range from 0 (worst performance) to 12 (best performance).
Change from baseline muscular strength by one repetition maximum test (1RM) | baseline, 20 days.
  1RM test for leg press is measured by kilograms. The one-repetition maximum (1RM) test is often considered as the 'gold standard' for assessing the strength capacity of individuals. It is simply defined as the maximal weight an individual can lift for only one repetition with correct technique.The 1RM machine leg press is often used as a measure of maximal lower body strength with older subjects.
Change from baseline grip strength by hydraulic hand dynamometer | baseline, 20 days.
  Grip muscle strength will be measured by kilograms.
Change from baseline balance parameters by Biodex Balance System SD | baseline, 20 days.
  Using Biodex Balance system with stable and unstable surface with open and closed eyes balance tests are performed (Limits of Stability, Fall Risk, Modified Clinical Test of Sensory Integration and Balance, Balance Error Scoring System).
Change from baseline stance and gait parameters by Zebris Medical GmbH | baseline, 20 days.
  Using Zebris medical GmbH platform stance and gait parameters are measured. It includes average forces for left and right foot, max load of body weight, foot rotation degree, Step length,Stride length,Step width,Stance, Swing and Double stance phases parameters, Step time,Stride time,Cadence,Velocity,Length of gait line,Single limb support line,Ant/post position,Lateral symmetry,Max gait line velocity,Force parameters, Load change, Maximum force, Maximum pressure,Time maximum force,Contact time.

SECONDARY OUTCOMES:
Change from baseline cardiopulmonary exercise capacity by maximal load (maxWatt) | baseline, 20 days.
  Maximal load measured with spiroergometry by maximal watts.
Change from baseline cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | baseline, 20 days.
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Raimondas Kubilius, prof, MD, Principal Investigator — LUHS hospital Kaunas Clinics Rehabilitation hospital of Kulautuva
Locations (1):
- LUHS hospital Kaunas Clinics Rehabilitation hospital of Kulautuva, Kaunas, Lithuania